CLINICAL TRIAL: NCT01693627
Title: Cemented Marathon/Corail Versus Pinnacle/Corail. Comparison of Polyethylene Wear, Component Migration and Periprosthetic Bone Mineral Density. A Randomised Study of 48 Hips Using Radiostereometry and Dual-energy X-ray Absorptiometry
Brief Title: Cemented Marathon/Corail Versus Pinnacle/Corail
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/133
Record Dates: First submitted 2012-03-21; First posted 2012-09-26 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Arthritis of the Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pinnacle/Corail with collar (Active Comparator): Uncemented THA using Pinnacle-100/Marathon XLPE(Depuy, Warsaw, IN) acetabular component and Corail(Depuy,Warsaw,IN)collared femoral stem with 32mm Alumina Biolox Forte(Depuy,Warsaw,IN). Tantalum beads will be inserted into periprosthetic bone.
  Interventions: Device: Pinnacle/Corail with collar
- Marathon/Corail with collar (Active Comparator): Reversed hybrid THA using cemented Marathon XLPE(Depuy,Warsaw,IN) acetabular component and an uncemented Corail(Depuy,Warsaw,IN)collared femoral component with 32 mm Alumina Biolox Forte(Depuy,Warsaw,IN)head. Tantalum beads will be inserted into periprosthetic bone.
  Interventions: Device: Marathon/Corail with collar
- Pinnacle/Corail without collar (Active Comparator): Uncemented THA using Pinnacle-100/Marathon XLPE(Depuy, Warsaw, IN) acetabular component and Corail(Depuy,Warsaw,IN)collarless femoral stem with 32mm Alumina Biolox Forte(Depuy,Warsaw,IN). Tantalum beads will be inserted into periprosthetic bone.
  Interventions: Device: Pinnacle/Corail without collar
- Marathon/Corail without collar (Active Comparator): Reversed hybrid total hip arthroplasty using cemented Marathon XLPE(Depuy,Warsaw,IN) acetabular component and an uncemented Corail(Depuy,Warsaw,IN)collarless femoral component with 32 mm Alumina Biolox Forte(Depuy,Warsaw,IN)head. Tantalum beads will be inserted into periprosthetic bone.
  Interventions: Device: Marathon/Corail without collar

INTERVENTIONS:
Device: Pinnacle/Corail with collar — Uncemented THA using Pinnacle-100/Marathon XLPE(Depuy, Warsaw, IN) acetabular component and Corail(Depuy,Warsaw,IN)collared femoral stem with 32mm Alumina Biolox Forte(Depuy,Warsaw,IN). Tantalum beads will be inserted into periprosthetic bone.
  Arms: Pinnacle/Corail with collar
Device: Marathon/Corail with collar — Reversed hybrid THA using cemented Marathon XLPE(Depuy,Warsaw,IN) acetabular component and an uncemented Corail(Depuy,Warsaw,IN)collared femoral component with 32 mm Alumina Biolox Forte(Depuy,Warsaw,IN)head. Tantalum beads will be inserted into periprosthetic bone.
  Arms: Marathon/Corail with collar
Device: Pinnacle/Corail without collar — Uncemented THA using Pinnacle-100/Marathon XLPE(Depuy, Warsaw, IN) acetabular component and Corail(Depuy,Warsaw,IN)collarless femoral stem with 32mm Alumina Biolox Forte(Depuy,Warsaw,IN). Tantalum beads will be inserted into periprosthetic bone.
  Arms: Pinnacle/Corail without collar
Device: Marathon/Corail without collar — Reversed hybrid total hip arthroplasty using cemented Marathon XLPE(Depuy,Warsaw,IN) acetabular component and an uncemented Corail(Depuy,Warsaw,IN)collarless femoral component with 32 mm Alumina Biolox Forte(Depuy,Warsaw,IN)head. Tantalum beads will be inserted into periprosthetic bone.
  Arms: Marathon/Corail without collar

SUMMARY:
A randomised, comparative, prospective, single-blinded trial of two hip prosthesis:

1. Marathon cemented all-poly acetabular cup(Depuy, Warsaw, Indiana), Corail uncemented femoral stem(Depuy, Warsaw, Indiana), 32mm Alumina Biolox Forte femoral head(Depuy, Warsaw, Indiana) and
2. Pinnacle/Marathon uncemented cup(Depuy, Warsaw, Indiana), Corail uncemented femoral stem(Depuy, Warsaw, Indiana), 32mm Alumina Biolox Forte femoral head(Depuy, Warsaw, Indiana)

There will be a further in-group randomisation to a Corail femoral stem with or without a collar, creating a number of 4 study-groups in total.

The aims of the study are:

* To compare polyethylene wear and migration of the moderately cross-linked Marathon polyethylene in a cemented version(Marathon) and in an uncemented cup(Pinnacle/Marathon)
* To evaluate micromigration and periacetabular bone mineral density of the 2 cups using radiostereometry(RSA)
* To evaluate the migration patterns and proximal femoral bone density changes around the Corail stems with and without a collar

ELIGIBILITY:
Inclusion Criteria:

* Age under 70 years with primary or secondary arthritis of the hip, aseptic necrosis of the femoral head, acute hip fracture or sequelae after hip fracture.

Exclusion Criteria:

* Active malignant disease, rheumatoid arthritis or other generalised auto-immune arthritic disease,
* BMI > 35,
* insulin dependent diabetes mellitus, 0 chronic or recurrent infection,
* liver disease,
* Paget's disease,
* dementia or lack of compliance for other reasons,
* uncompensated cardiac or pulmonary disease(ASA class 3 or 4). Prosthesis in the contralateral hip does not exclude the patient, but only one hip in each patient can be included in the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-01; Primary Completion 2017-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Polyethylene wear | After 5 years of follow-up
  Comparison of polyethylene wear rates in a modular uncemented acetabular component and a cemented all-polyethylene acetabular component using radiostereometric analysis
Component migration-cup | After 5 years of follow-up
  Comparison of the migration of a modular uncemented acetabular component and a cemented all-polyethylene acetabular component using radiostereometric analysis.
Periprosthetic bone mineral density | After 2 years of follow-up
  Differences in bone mineral density around a cemented and an uncemented acetabular component using Dual X-ray absorptiometry. Differences in bone mineral density around an uncemented fully HA-coated femoral component with or without a collar using Dual X-ray absorptiometry.
Component migration-stem | After 5 years of follow-up
  Comparison of the migration of an uncemented fully HA-coated femoral component with and without a collar using radiostereometric analysis.

SECONDARY OUTCOMES:
Clinical outcome | After 5 years of follow-up
  Comparison of clinical results between study groups using HHS and PROMs

CONTACTS AND LOCATIONS:
Overall Officials: Leif I Havelin, MD, PhD, Study Director — Department of Orthopeadic Surgery, Haukeland University Hospital, Bergen, Norway; Benedikt A Jonsson, MD, Principal Investigator — Department of Orthopeadic Surgery, Haukeland University Hospital, Bergen, Norway; Geir Hallan, MD, PhD, Principal Investigator — Department of Orthopeadic Surgery, Haukeland University Hospital, Bergen, Norway; Ove Furnes, MD, PhD, Study Chair — Department of Orthopeadic Surgery, Haukeland University Hospital, Bergen, Norway; Clara G Gjesdal, MD, PhD, Study Chair — Department of Rheumatology, Haukeland University Hospital, Bergen, Norway; Kristin Haugan, MA, Study Chair — Department of Orthopeadic Surgery, Trondheim University Hospital, Trondheim, Norway; Arne K Skredderstuen, MD, Study Chair — Department of Orthopeadic Surgery, Haukeland University Hospital, Bergen, Norway; Terje Stokke, Study Chair — Department of Radiology, Haukeland University Hospital, Bergen, Norway
Locations (1):
- Department of Orthopaedic Surgery, Haukeland University Hospital, Bergen, Norway